

# Statistical Analysis Plan (SAP)

KIC-START: A low-interventional, prospective, multi-center study to evaluate real-world clinical, biochemical and patient-reported responses to tofacitinib induction therapy in patients with moderately to severely active ulcerative colitis in Switzerland

# **Administrative Information**

| Project number: | 1594 |
|----------------------------|------------------------------------------|
| Trial registration number: | A3921395; clinicaltrials.gov NCT05069259 |
| SAP version: | SAP version 1.0 (31 July 2024) |
| Protocol version: | Final Protocol, 22 March 2022 |

| CTU Bern SAP for: Study A3921395 KIC-START | | Version: 1.0 | |
|---|---|---|---|
| | T | \(\(\text{i}\) = 00 | |
| CTU Bern | Template: Statistical Analysis Plan (SAP) | Version: 03 | Dogo 4 of 44 |



Faculty of Medicine CTU Bern

# Contributors

| Name | Affiliation | Role in SAP writing |
|------|-------------|---------------------|
| PPD | CTU Bern | Author |
| PPD | CTU Bern | Author |

# **Revision history**

| Revision | Justification | Timing |
|----------|---------------|--------|

# Approved by

| Name | Affiliation | Study Role | Date and Signature |
|------|-------------|---------------------|--------------------|
| PPD | CTU Bern | Trial Statistician | PPD |
| PPD | CTU Bern | Senior Statistician | PPD |
| PPD | Pfizer Inc. | Study Statistician | PPD |

|----------|-------------------------------------------|--------------|
| | Tourists Objects I Apply in DirectOAD | 1/ |
| CTU Bern | Template: Statistical Analysis Plan (SAP) | Version: 03 |

Valid from: 28.02.2019


Code: CS\_STA\_TEM-11





# 1. Glossary of abbreviations

Code: CS\_STA\_TEM-11

| CRF | Case Report Form |
|-------|--------------------------------------------|
| EDC | Electronic Data Capturing system |
| FAS | Full Analysis Set |
| fCAL | Fecal calprotectin |
| IBDQ | Inflammatory Bowel Disease Quality of Life |
| ICD | Informed Consent Document |
| IUS | Intestinal Ultrasound |
| OTAS | On-Tofacitinib Analysis Set |
| PMS | Partial Mayo Score |
| PP | Per-Protocol analysis set |
| PRO | Patient-Reported Outcome |
| (S)AE | Serious Adverse Event |
| SOC | System Organ Class |
| SOP | Standard Operating Procedure |
| UC | Ulcerative Colitis |
| W | Week |

|-----------|-------------------------------------------|--------------|
| CTU Barra | Template: Statistical Analysis Plan (SAP) | Version: 03 |
| CTU Bern | | |

Valid from: 28.02.2019

Page **3** of **44** 



Faculty of Medicine
CTU Bern

# Contents

| 1. | Glos | ssary of abbreviations | | 3 |
|---|---|---|---|---|
| 2. | Intro | oduction | | 7 |
| 2.1 | Bac | kground and rationale | | 7 |
| 2.2 | Obje | ectives | | 7 |
| 3. | Stud | dy methods | | 8 |
| 3.1 | Tria | I design | | 8 |
| 3.2 | Ran | domization | | 8 |
| 3.3 | Sam | ple size | | 8 |
| 3.4 | Frar | nework | | 8 |
| 3.5 | Stat | istical interim analyses and stopping guida | ance | 8 |
| 3.6 | Timi | ing of final analysis | | 8 |
| 3.7 | Timi | ing of outcome assessments | | 8 |
| 3.8 | Bline | ding | | 8 |
| 4. | Data | a management | | 9 |
| 4.1 | Data | a export | | 9 |
| 4.2 | Data | a validation | | 9 |
| 4.3 | Data | a preparation | | 9 |
| 5. | Stat | istical principles | | 15 |
| 5.1 | Con | fidence intervals and P values | | 15 |
| 5.2 | Ana | lysis populations | | 15 |
| 5.2.1 | Full | analysis set (FAS) | | 15 |
| 5.2.2 | Per- | protocol analysis set (PP) | | 15 |
| 5.2.3 | On-1 | tofacitinib analysis set (OTAS) | | 15 |
| CTU Be | ern | SAP for: Study A3921395 KIC-START | Version: 1.0 | |
| | - | Template: Statistical Analysis Plan (SAP) | Version: 03 | |
| CTU Beri | 'n | Code: CS_STA_TEM-11 | Valid from: 28.02.2019 | Page <b>4</b> of <b>44</b> |



| 5.2.4 | Safety population | | 15 |
|---|---|---|---|
| 6. | Study Population | | 16 |
| 6.1 | Screening data | | 16 |
| 6.2 | Eligibility | | 16 |
| 6.2.1 | Inclusion Criteria | | 16 |
| 6.2.2 | Exclusion Criteria | | 16 |
| 6.3 | Recruitment | | 17 |
| 6.4 | Baseline patient characteristics | | 18 |
| 6.5 | Procedural characteristics (if applicable) | | 24 |
| 6.6 | Adherence and protocol deviations | | 24 |
| 6.7 | Withdrawal/follow-up | | 24 |
| 7. | Analysis | | 25 |
| 7.1 | Outcome definitions | | 25 |
| 7.2 | Analysis methods | | |
| 7.2.1 | Primary analysis | | |
| 7.2.2 | Secondary analyses | | |
| 7.2.3 | Sensitivity analyses | | |
| 7.2.4 | Subgroup analyses | | |
| 7.2.5 | Additional analyses | | |
| 7.3 | Interim analyses | | |
| 7.4 | Missing data | | |
| 7.5 | Safety evaluation | | |
| 7.6 | Subproject (if applicable) | | |
| 7.7 | Statistical software | | |
| 7.8 | Quality control | | |
| СТИ В | ern SAP for: Study A3921395 KIC-START | Version: 1.0 | |
| | Template: Statistical Analysis Plan (SAP) | Version: 03 | |
| CTU Be | Code: CS_STA_TEM-11 | Valid from: 28.02.2019 | Page <b>5</b> of <b>44</b> |



| 8. | Presentation of the results - Tables, Listings and Figures | 35 |
|---|---|---|
| 8.1 | Figures | 35 |
| 8.1.1 | Flow chart | 35 |
| 8.1.2 | Course of the PMS, PROs and fCAL concentration. | 36 |
| 8.2 | Tables | 36 |
| 8.2.1 | Study participants | 36 |
| 8.2.2 | Efficacy Outcomes at W8 and W16 | 37 |
| 8.2.3 | Temporal variation of PMS, PROs and fCAL concentration | 38 |
| 8.3 | Correlation between PRO and PMS, IBDQ score and fCAL concentrations outcomes | 40 |
| 8.4 | Additional exploratory outcomes | 41 |
| 8.5 | Safety Data | 42 |
| 8.5.1 | Summary of AEs | 42 |
| 8.5.2 | Severity of AEs, by system organ class and preferred term | 42 |
| 9. | Changes from the protocol | 43 |
| 10. | References | 44 |

|---|---|---|
| Code: CS_STA_TEM-11 | Valid from: 28.02.2019 | Page <b>6</b> of <b>44</b> |



### 2. Introduction

### 2.1 Background and rationale

A number of studies have been published demonstrating tofacitinib's safety and efficacy profile in ulcerative colitis (UC) [1-8]. While it is known that tofacitinib therapy is associated with a rapid onset of symptom relief in terms of the Partial Mayo score (PMS) components (stool frequency and rectal bleeding), the response of other important patient-reported outcomes (PROs), such as fatigue, urgency and abdominal pain, are less well characterized [9, 10]. Measuring these PROs will provide a broader understanding of how patients experience response to tofacitinib treatment. Moreover, the response of intestinal inflammation to tofacitinib induction therapy is currently not fully understood [11]. Regular measurements of fecal calprotectin (fCAL) levels, a widely used biomarker in UC, will provide a measure of the response of intestinal inflammation to tofacitinib treatment. Early measurements will assess the validity of fCAL as an early biochemical predictor of treatment response.

#### 2.2 Objectives

This study aims to generate granular real-world data on tofacitinib therapy in UC and enable a characterization of the relationship between changes in PMS, PROs and intestinal inflammation during tofacitinib induction therapy.

| CTU Bern SAP for: Study A3921395 KIC-START Version: 1.0 | | Version: 1.0 | |
|---|---|---|---|
| | Code: CS STA TEM-11 | Valid from: 28.02.2019 | Page <b>7</b> of <b>44</b> |



# 3. Study methods

### 3.1 Trial design

This study is a single-arm, open-label, prospective, low-interventional, multi-center study conducted in Switzerland in a real-world setting without any comparison groups. Approximately 60 participants were planned to be enrolled. However, following the termination decision as per Pfizer CT26-GSOP, recruitment was prematurely stopped after the enrollment of 18 patients. Please see Section 9 for details on the resulting changes to endpoints and analysis specified in the protocol.

#### 3.2 Randomization

Not applicable.

# 3.3 Sample size

The initial sample size calculation was shown in the final version of the protocol (22 March 2022). According to that calculation, a total of approximately 60 participants were planned to be enrolled into the study. However, following an internal decision by Pfizer, recruitment was prematurely stopped after the enrollment of 18 patients.

We expect that 60% of participants will achieve a clinical response at Week 8. As noted in the protocol, a sample of 60 participants would have result in a 2-sided 95% Wilson confidence interval around a frequency of 60% from 47.4 to 71.4%. A sample of 18 participants will result in a 2-sided 95% Wilson confidence interval around a frequency of 60% from 37.6 to 78.9%.

#### 3.4 Framework

This is a descriptive single-arm study, there will be no formal hypothesis testing.

#### 3.5 Statistical interim analyses and stopping guidance

Not applicable.

#### 3.6 Timing of final analysis

Final analysis will be performed after database lock.

#### 3.7 Timing of outcome assessments

All outcomes will be analyzed collectively after study completion. After completion of data entry, data validation and cleaning will be performed. Data analysis will start after database lock.

### 3.8 Blinding

The study is unblinded.

| CTU Bern SAP for: Study A3921395 KIC-START Version: 1.0 | | Version: 1.0 | |
|---|---|---|---|
| | 1 | | |
| C LO Delli | O OO OTA TEM 44 | \/-!:-! f 00 00 0040 | Dama 0 of 44 |



# 4. Data management

# 4.1 Data export

The Data Management system used in this study is a dedicated electronic data capturing (EDC) system, secuTrial. The EDC system is activated for the study only once a formal test procedure has been passed successfully. All data entered in the EDC system are stored on a Linux server in a dedicated Oracle database at Inselspital Bern, Switzerland.

Clinical study data will be provided by CTU Bern (Clinical Trial Unit of the University of Bern) in a data-base format (secuTrial®) and will be imported into R by the study statistician for data preparation, validation, and analysis.

#### 4.2 Data validation

First line data validation is performed by the online Case Report Form (eCRF) system in real-time as defined in the data dictionary. Second line data validation and cleaning will be performed according to the Standard Operating Procedure (SOP) for data validation [13] after the completion of overall data collection, before database export for the final analysis.

### 4.3 Data preparation

Table 4-a: Data preparation

| Variable definition | Variable type | Derivation |
|---|---|---|
| Baseline date: date of first medication intake | Date (dd.mm.yyyy) | pro_medi_start_date |
| Prior exposure to TNFi, vedolizumab and ustekinumab; | Binary (yes, no) | Used variables: th_ustekinumab th_vedolizumab th_tnfi Visit: Baseline. Derivation - General: 'yes' if at least one of the above variables is different from 'Never prescribed'; 'No' otherwise if missing data (i.e., at least one of the 3 variables mentioned above is missing): 'yes' if at least one of the above variables is different from "Never prescribed"; 'NA' otherwise. |
| Concomitant medication with corticosteroids or aminosalicylic acids | Binary (yes, no) | Used variables: cm_drug.factor cm_start cm_end pro_medi_start_date Derivation If cm_drug.factor contains "Topical corticosteroids" OR "Oral corticosteroids" OR "Topical aminosalicylates" OR "Oral aminosalicylates" |

|---|---|---|---|
| OTU D | Template: Statistical Analysis Plan (SAP) | Version: 03 | |
| CTU Bern | Code: CS STA TEM-11 | Valid from: 28.02.2019 | Page <b>9</b> of <b>44</b> |



b UNIVERSITÄT BERN

Faculty of Medicine

CTU Bern

| Variable definition | Variable type | Derivation |
|---|---|---|
| | | AND if one of the mentioned above drugs is taken at the pro_medi_start_date (i.e. pro_medi_start_date %in% [cm_start, cm_end]) |
| Concomitant use of Ustekinumab | Binary (yes, no) | Used variables: cm_drug.factor cm_start cm_end pro_medi_start_date Derivation If cm_drug.factor contains "Ustekinumab" AND if one of the mentioned above drugs is taken at the pro_medi_start_date (i.e. pro_medi_start_date %in% [cm_start, cm_end]) |
| Concomitant use of Vedolizumab | Binary (yes, no) | Used variables: cm_drug.factor cm_start cm_end pro_medi_start_date Derivation If cm_drug.factor contains "Vedolizumab" AND if one of the mentioned above drugs is taken at the pro_medi_start_date (i.e. pro_medi_start_date %in% [cm_start, cm_end]) |
| Concomitant use of TNF inhibitors | Binary (yes, no) | Used variables: cm_drug.factor cm_start cm_end pro_medi_start_date Derivation If cm_drug.factor contains "TNF inhibitors" AND if one of the mentioned above drugs is taken at the pro_medi_start_date (i.e. pro_medi_start_date %in% [cm_start, cm_end]) |
| Concomitant use of Tacrolimus | Binary (yes, no) | Used variables: cm_drug.factor cm_start cm_end pro_medi_start_date Derivation If cm_drug.factor contains "Tacrolimus" AND if one of the mentioned above drugs is taken at the pro_medi_start_date (i.e. pro_medi_start_date %in% [cm_start, cm_end]) |
| Concomitant use of Cyclosporin | Binary (yes, no) | Used variables: cm_drug.factor cm_start cm_end pro_medi_start_date Derivation If cm_drug.factor contains "Cyclosporin" AND if one of the mentioned above drugs is taken at the pro_medi_start_date (i.e. pro_medi_start_date %in% [cm_start, cm_end]) |
| Concomitant use of Methotrexate | Binary (yes, no) | Used variables: cm_drug.factor cm_start cm_end pro medi start date |

| OTIL D. | Template: Statistical Analysis Plan (SAP) | Version: 03 |
|---|---|---|
| CTU Bern | Code: CS_STA_TEM_11 | Valid from: 28 02 2019 |

Version: 1.0

SAP for: Study A3921395 KIC-START



Faculty of Medicine

CTU Bern

| Variable definition | Variable type | Derivation |
|---|---|---|
| | | Derivation If cm_drug.factor contains "Methotrexate" AND if one of the mentioned above drugs is taken at the pro_medi_start_date (i.e. pro_medi_start_date %in% [cm_start, cm_end]) |
| Concomitant use of Thiopurines | Binary (yes, no) | Used variables: cm_drug.factor cm_start cm_end pro_medi_start_date Derivation If cm_drug.factor contains "Thiopurines" AND if one of the mentioned above drugs is taken at the pro_medi_start_date (i.e. pro_medi_start_date %in% [cm_start, cm_end]) |
| Concomitant use of aminosalicy-lates | Binary (yes, no) | Used variables: cm_drug.factor cm_start cm_end pro_medi_start_date Derivation If cm_drug.factor contains "Oral / topical aminosalicylates" AND if one of the mentioned above drugs is taken at the pro_medi_start_date (i.e. pro_medi_start_date %in% [cm_start, cm_end]) |
| Concomitant use of steroids | Binary (yes, no) | Used variables: cm_drug.factor cm_start cm_end pro_medi_start_date Derivation If cm_drug.factor contains "Topical corticosteroids" OR "Oral corticosteroids" AND if one of the mentioned above drugs is taken at the pro_medi_start_date (i.e. pro_medi_start_date %in% [cm_start, cm_end]) |
| Concomitant use of low dose steroids | Binary (yes, no) | Used variables: cm_drug.factor cm_start cm_end pro_medi_start_date cm_dose Derivation If cm_drug.factor contains "Topical corticosteroids" OR "Oral corticosteroids" AND if one of the mentioned above drugs is taken at the pro_medi_start_date (i.e. pro_medi_start_date %in% [cm_start, cm_end]) with the dose (i.e. cm_dose) %in% c( 'Systemic: < 15mg/day prednisone equivalent', 'Locally- acting: < 3mg/day budesonide') |
| Concomitant use of high dose steroids | Binary (yes, no) | Used variables: cm_drug.factor cm_start cm_end pro_medi_start_date cm_dose Derivation If cm_drug.factor contains "Topical corticosteroids" OR |

|---|--------------------------------------------|---|--------------|
| | • | | |
| ſ | | T | 1/ : 00 |

| CTU Barra | Template: Statistical Analysis Plan (SAP) | Version: 03 | |
|---|---|---|---|
| CTU Bern | Code: CS_STA_TEM-11 | Valid from: 28.02.2019 | Page <b>11</b> of <b>44</b> |



Faculty of Medicine

CTU Bern

| Variable definition | Variable type | Derivation |
|---|---|---|
| | | "Oral corticosteroids" AND if one of the mentioned above drugs is taken at the pro_medi_start_date (i.e. pro_medi_start_date %in% [cm_start, cm_end]) with the dose (i.e. cm_dose) %in% c( 'Systemic: ≥ 15mg/day prednisone equivalent', 'Locallyacting: ≥ 3mg/day budesonide') |
| Baseline predominant tofacitinib dose | Binary (<15mg tofacitinib/day, ≥15 mg tofacitinib/day) | Variable: te_bl_dose.factor te_bl_dose_oth_value te_bl_dose_oth_unit Visit: Baseline. Derivation 'yes' if te_bl_dose.factor == '10 mg twice daily' OR |
| | | <pre>te_bl_dose.factor == 'Other' &amp; (te_bl_dose_oth_value &amp; te_bl_dose_oth_unit &lt;15 mg/day); otherwise 'no'.</pre> |
| Average daily dose of Tofacitinib during the trial | Binary (<15mg tofa-<br>citinib/day, ≥15 mg tofa-<br>citinib/day) | Variable: te_bl_dose.factor te_bl_dose_oth_value te_bl_dose_oth_unit te_dose te_other_value te_other_unit te_start te_end te_disc_date Derivation: Calculation of the mean daily dose of tofacitinib and categorization as < 15mg/day or ≥ 15mg/day |
| IBDQ score | Continuous (score varying between from 32 to 224) | Variables: pro_ibdq_x (with X varying from 1 to 32) Derivation: at each reported time point. For each variable, 7 answers are possible. Answers are ranked from the 'worst' to 'best' quality of life, and replaced by a score varying from 1(worst) to 7(best). Scores obtained for each of the 32 variables are then summed up. If any of the pro_ibdq_x (with X varying from 1 to 32) variables is missing the score is coded as missing. |
| Weekly fatigue score (FACIT-F score) | Continuous (score varying between from 0 to 52) | Variables pro_facit_an1, pro_facit_an2, pro_facit_an3, pro_facit_an4, pro_facit_an5, pro_facit_an7, pro_facit_an8, pro_facit_an12, pro_facit_an14, pro_facit_an15, pro_facit_an16, pro_facit_hi12, pro_facit_hi7 Derivation: at each reported time point. For each variable, 5 answers are possible. Answers are converted to score (see below), scores obtained for each of the 13 listed variables are then summed up. If any of the variables use to derive the score is missing the score is coded as missing. |
| CTU Bern SAP for: Study A39 | 1<br>121395 KIC-START | Version: 1.0 |
| | | 1 |

| OTU Dama | Template: Statistical Analysis Plan (SAP) | Version: 03 | |
|---|---|---|---|
| CTU Bern | Code: CS_STA_TEM-11 | Valid from: 28.02.2019 | Page <b>12</b> of <b>44</b> |



Faculty of Medicine

CTU Bern

| Variable defini | tion | Variable type | Derivation |
|---|---|---|---|
| | | | Scoring system: |
| | | | Not at all =0; A little bit =1; Somewhat =2; Quite a bit =3; Very much =4 |
| PMS score | | Continuous | Variables: pms_stool_freq, pms_rect_bleed, pms_glob_ass Derivation: At each reported time point. For each variable, 4 answers are possible. Answers are converted to score from 0 (nor- mal) to 3 (more severe condition), scores obtained for each of the 3 listed variables are then summed up. If any of the variables use to derive the score is missing the score is coded as missing. |
| PMS stool frequency subscore | | Continuous | Variable: pms_stool_freq Derivation: At each reported time point. 4 answers are possible. Answers are converted to score from 0 (normal) to 3 (more severe condition). |
| PMS rectal bleeding subscore | | Continuous | Variable: pms_rect_bleed Derivation: At each reported time point. 4 answers are possible. Answers are converted to score from 0 (normal) to 3 (more severe condition). |
| PMS physician's global assessment subscore | | Continuous | Variable: pms_glob_ass Derivation: At each reported time point. 4 answers are possible. Answers are converted to score from 0 (normal) to 3 (more severe condition). |
| Full Mayo score | | Continuous | Variables: PMS score (see above), ra_mayo_subscore Derivation: At each reported time point. For each variable, 4 answers are possible for the ra_mayo_subscore variable. Answers are converted to score from 0 (normal) to 3 (severe disease), scores obtained for the PMS score and the ra_mayo_subscore variable are then summed up. If any of the variables use to derive the score is missing the score is coded as missing. |
| Participant's age | | Continuous | Used variables: ic_date, ymob Derivation: Date of signature of the inform consent in mm.yyyy – the date of birth in mm.yy. Result is given in year and rounded to one decimal point |
| EIM improvement status at week_x (x can be equal to 8 or 16) | | Continuous | Variables: eim_cat, eim_subcat_muco, eim_subcat_muscu, eim_subcat_ocular, eim_subcat_hepa, eim_ac- tivity Derivation: For each EIM (defined by the variables eim_cat, eim_subcat_muco, eim_subcat_muscu, eim_sub- cat_ocular, eim_subcat_hepa) •'No worsening' if |

 CTU Bern
 Template: Statistical Analysis Plan (SAP)
 Version: 03

 Code: CS\_STA\_TEM-11
 Valid from: 28.02.2019
 



Faculty of Medicine

CTU Bern

| Variable definition | Variable type | Derivation |
|---|---|---|
| | | eim_activity at baseline =' Active at assessment' AND eim_activity at week_x =' Active at assessment' OR eim_activity at baseline =' Past, but not active' AND eim_activity at week_x =' Past, but not active' OR EIM at baseline AND EIM not mentionned at week_x ='Worsened' if eim_activity at baseline =' Past, but not active' AND eim_activity at week_x =' Active at assessment' ='Improved' if eim_activity at baseline =' Active at assessment' AND eim_activity at week_x =' Past, but not active' ='New occurence' if No EIM at baseline AND eim_activity at week_x =' Active at assessment' |
| Number of comorbidities | Continuous | Used variables: co_morb_yn co_morb Derivation: at bl, W8 and 16. If co_morb_yn== 'yes' count the number of different entries for co_morb If co_morb_yn== 'no' 0 |
| Number of EIMs | Continuous | Used variables: eim_yn Derivation: at bl, W8 and 16. If eim_yn== 'yes' count the number of different entries for EIM If eim_yn== 'no' 0 |
| uMARS score | Continuous | Sum all uMARS answers (variables names not available at the time of writing the SAP). If any of the variables use to derive the score is missing, the score is coded as missing. |

|---|---|---|---|
| CTIL Bown | Template: Statistical Analysis Plan (SAP) | Version: 03 | |
| CTU Bern | Code: CS_STA_TEM-11 | Valid from: 28.02.2019 | Page <b>14</b> of <b>44</b> |



# 5. Statistical principles

### 5.1 Confidence intervals and P values

All confidence intervals will be two-sided and relate to the 95% level and the two-sided significance level will be set at  $\alpha = 0.05$ .

### 5.2 Analysis populations

# 5.2.1 Full analysis set (FAS)

The full analysis set (FAS), will include all participants who were included in the study (i.e., performed baseline visit and received a study identification number). This analysis will therefore include all study participants, regardless of their adherence to study protocol procedures.

### 5.2.2 Per-protocol analysis set (PP)

Not applicable.

# 5.2.3 On-tofacitinib analysis set (OTAS)

The on-tofacitinib analysis set consists of all participants in the FAS set who did not stop or interrupt the tofacitinib therapy before the 8 weeks visit.

Table 5-a: Derivation of protocol deviations

| Protocol deviation | eCRF sheet | Variable | Variable type | Derivation |
|---|---|---|---|---|
| Completion of the therapy until the W8 visit | Binary (yes, no) | Used variables: Time to tofacitinib discontinuation (see above) Date of the 8 weeks visit Derivation 'yes' if Time to tofacitinib discontinuation (see above) < Date of the 8 weeks visit | Completion of<br>the therapy until<br>the W8 visit | Binary (yes, no) |

# 5.2.4 Safety population

Not applicable

|-------------------------------------------|--------------|
| Tampleto: Statistical Analysis Plan (SAR) | Vargion: 03 |

|---|---|---|---|
| CTU Bern | Code: CS_STA_TEM-11 | Valid from: 28.02.2019 | Page <b>15</b> of <b>44</b> |



# 6. Study Population

### 6.1 Screening data

All screening evaluations will be entered in the database. In case of screening failure, reason(s) for failure will be recorded.

### 6.2 Eligibility

#### 6.2.1 Inclusion Criteria

### Age and Sex:

Male or female participants 18 years of age or older at screening visit;

### Type of Participant and Disease Characteristics:

- Participants with confirmed diagnosis of UC and who are prescribed tofacitinib (Xeljanz®) for moderately to severely active UC as per the Swiss label [14] and as per physician's clinical judgement, independently of this study;
- Participants who are willing and able to comply with all scheduled visits, treatment plan, study interventions (Section 6 of the protocol), and other study procedures (Section 8 of the protocol).

#### Informed Consent:

 Capable of giving personally signed informed consent (as described in Section 10.1.4 of the protocol), which includes compliance with the requirements and restrictions listed in the Informed Consent Form (ICD) and in the protocol.

#### 6.2.2 Exclusion Criteria

#### **Medical Conditions:**

Presence of clinical findings suggestive of Crohn's disease;

#### **Prior/Concomitant Therapy:**

- Any previous exposure to tofacitinib including participation in the tofacitinib clinical program;
- Co-medication with any other advanced therapies for UC (biologics\*, azathioprine, mercaptopurine and methotrexate) or any other JAK inhibitor.
  - \*TNF, integrin or cytokine antagonists.

#### Other Exclusions:

- Any identified contra-indications for use of tofacitinib as per the Swiss label [14];
- Not owning a handheld digital device compatible with the Sidekick Health App, not willing to have it installed on this device or not capable of using the App;
- Investigator site staff or Pfizer employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family members.

| CTU Ber | SAP for: Study A3921395 KIC-START | Version: 1.0 | |
|---|---|---|---|
| CTU Barr | Template: Statistical Analysis Plan (SAP) | Version: 03 | |
| CTU Berr | | Valid from: 28 02 2019 | Page <b>16</b> of <b>44</b> |



#### 6.3 Recruitment

A CONSORT patient flow diagram will be drawn following the CONSORT 2010 standards [15].



|---|---|---|
| Code: CS STA TEM-11 | Valid from: 28.02.2019 | Page <b>17</b> of <b>44</b> |



# 6.4 Baseline patient characteristics

The patient characteristics at baseline will be presented in a table, as number and percentage or mean and standard deviation for categorical and normally distributed continuous variables, respectively. For data severely deviating from a normal distribution, we will present median and quartiles.

Table 6-a: Baseline table

| Description | Variable | Туре |
|---|---|---|
| Patient demographic | Patient demographics | |
| Age (year of birth) | ic_date and ymob (see data preparation 4.3) | Continuous: years |
| Gender | sex | Binary: Male, Female |
| ВМІ | dg_bmi | Continuous |
| Smoking status | dg_smoking | Categorical: Never smoked, Former smoker,<br>Current smoker |
| Concomitant medica | ation at baseline | |
| Concomitant medication with corticosteroids or aminosalicylic acids | see data preparation 4.3 | Binary: Yes, No |
| <ul> <li>Concomitant use<br/>of steroids</li> </ul> | see data preparation 4.3 | |
| <ul> <li>Concomitant use<br/>of low dose steroids</li> </ul> | see data preparation 4.3 | |
| <ul> <li>Concomitant use<br/>of high dose ster-<br/>oids</li> </ul> | see data preparation 4.3 | Binary: Yes, No |
| Concomitant use of<br>Ustekinumab | see data preparation 4.3 | Binary: Yes, No |
| Concomitant use of<br>Vedolizumab | see data preparation 4.3 | Binary: Yes, No |
| Concomitant use of TNF inhibitors | see data preparation 4.3 | Binary: Yes, No |
| Concomitant use of<br>Tacrolimus | see data preparation 4.3 | Binary: Yes, No |
| Concomitant use of Cyclosporin | see data preparation 4.3 | Binary: Yes, No |
| Concomitant use of<br>Methotrexate | see data preparation 4.3 | Binary: Yes, No |
| Concomitant use of Thiopurines | see data preparation 4.3 | Binary: Yes, No |
| Concomitant use of aminosalicylates | see data preparation 4.3 | Binary: Yes, No |
| UC medication | | |

|---|---|---|---|
| OTU D | Template: Statistical Analysis Plan (SAP) | Version: 03 | |
| CTU Bern | Code: CS_STA_TEM-11 | Valid from: 28.02.2019 | Page <b>18</b> of <b>44</b> |



| Description | Variable | Туре |
|---|---|---|
| Baseline<br>predominant<br>tofacitinib dose | see data preparation 4.3 | Binary: < 15mg; or ≥ 15mg to facitinib/day |
| Main UC disease cha | aracteristics | |
| PMS | see data preparation 4.3 | Continuous |
| PMS stool frequency subscore | see data preparation 4.3 | Continuous |
| PMS rectal bleeding subscore | see data preparation 4.3 | Continuous |
| PMS physician's global assessment subscore | see data preparation 4.3 | Continuous |
| UC treatment history | 1 | |
| Prior exposure to TNFi,vedolizumab and ustekinumab | th_ustekinumab, th_vedolizumab, and th_tnfi at baseline (see data preparation 4.3) | Binary: Yes, No |
| Prior exposure to TNFi | th_tnfi_nr at baseline ('no' if th_tnfi_nr = 'Never prescribed', 'yes' otherwise) | Binary: Yes, No |
| □ Number of TNFi □ Number o | th_tnfi_nr | Binary: 1, >1 |
| <ul> <li>Prior exposure to<br/>oral &amp; topical ami-<br/>nosalicylates</li> </ul> | th_amino | Categorical: Never prescribed, Lack of/ insufficient response, Loss of response, Intolerance/side effects, Treatment ongoing, Unknown |
| <ul> <li>Prior exposure to<br/>Locally acting &amp; sys-<br/>temic corticosteroids<br/>(e.g. budesonide,<br/>prednisone)</li> </ul> | th_cortico | Categorical: Never prescribed, Lack of/ insufficient response, Loss of response, Intolerance/side effects, Treatment ongoing, Unknown |
| <ul> <li>Prior exposure to<br/>Thiopurines (e.g.<br/>AZA, 6-MP)</li> </ul> | th_thiopur | Categorical: Never prescribed, Lack of/ insufficient response, Loss of response, Intolerance/side effects, Treatment ongoing, Unknown |
| <ul> <li>Prior exposure to<br/>Other immunosup-<br/>pressants (e.g. cy-<br/>closporine, tacroli-<br/>mus)</li> </ul> | th_immunosup | Categorical: Never prescribed, Lack of/ insufficient response, Loss of response, Intolerance/side effects, Treatment ongoing, Unknown |
| □ Prior exposure to<br>TNF inhibitors<br>(TNFi) | th_tnfi | Categorical: Never prescribed, Lack of/ insufficient response, Loss of response, Intolerance/side effects, Treatment ongoing, Unknown |
| Prior exposure to vedolizumab | th_vedolizumab at baseline ('no' if th_vedoli-<br>zumab = 'Never prescribed', 'yes' otherwise) | Binary: Yes, No |

|---|---|---|---|
| CTU Bown | Template: Statistical Analysis Plan (SAP) | Version: 03 | |
| CTU Bern | Code: CS_STA_TEM-11 | Valid from: 28.02.2019 | Page <b>19</b> of <b>44</b> |



| Description | Variable | Туре |
|---|---|---|
| Prior exposure to ustekinumab | th_ustekinumab at baseline ('no' if th_ustekinumab = 'Never prescribed', 'yes' otherwise) | Binary: Yes, No |
| Prior exposure to oral & topical aminosalicylates | th_amino at baseline ('no' if th_amino = 'Never prescribed', 'yes' otherwise) | Binary: Yes, No |
| Prior exposure to lo-<br>cally acting & sys-<br>temic corticosteroids<br>(e.g. budesonide,<br>prednisone) | th_cortico at baseline ('no' if th_cortico = 'Never prescribed', 'yes' otherwise) | Binary: Yes, No |
| Prior exposure to Thiopurines (e.g. AZA, 6-MP) | th_thiopur at baseline ('no' if th_thiopur = 'Never prescribed', 'yes' otherwise) | Binary: Yes, No |
| Prior exposure to IMP | th_imp at baseline ('no' if th_imp_yesno="no" OR th_imp = 'Never prescribed', 'yes' otherwise) | Binary: Yes, No |
| Prior exposure to other treatment | th_imp at baseline ('no' if th_other_yesno<br>="no" OR th_other = 'Never prescribed', 'yes'<br>otherwise) | Binary: Yes, No |
| Other immunosup-<br>pressants (e.g. cy-<br>closporine, tacroli-<br>mus) | th_immunosup | |
| SOC Intestinal Ultra | Sound (IUS) | |
| For Ascending, descending, Sigmoid and transverse colon at W8 & 16 | <pre>ra_[*]_col_ext [*] = - 'asc' for Ascending colon</pre> | Binary: Yes, no |
| Extension of wall-<br>thickening | - 'desc' for descending colon - 'sig' for Sigmoid colon - 'trans' for transverse colon | 2a.y. 7 ee, 1.e |
| For Ascending, descending, Sigmoid and transverse colon at W8 & 16 Normalization of wall-thickening | ra_[*]_col_norm [*] = - 'asc' for Ascending colon - 'desc' for descending colon - 'sig' for Sigmoid colon - 'trans' for transverse colon | Binary: Yes, no |
| Loss of stratification at W8 & 16 | ra_loss_strat | Binary: Yes, no |
| Loss of colonic<br>haustration at W8 &<br>16 | ra_loss_col_haus | Binary: Yes, no |

|---|---|---|
| C TO Delli | Code: CS_STA_TEM-11 | Valid from: 28 02 2019 |



| Description | Variable | Туре |
|---|---|---|
| Structure formation at W8 & 16 | ra_struct_form | Binary: Yes, no |
| Hyperechogenic re-<br>action adjacent to<br>the bowel wall | ra_hyper_react | Binary: Yes, no |
| Co-morbidities, inclu | uding extra-intestinal manifestations | |
| Co-morbidities | | |
| Number of comorbidities | see data preparation 4.3 | Continuous |
| Extraintestinal Mani | festations (EIM) | |
| Identified EIM | eim_yn | Binary: yes, no |
| Number of EIMs | see data preparation 4.3 | Continuous |
| Mucocutaneous | <pre>eim_cat ('yes' if eim_cat = 'Mucocutaneous', 'no' otherwise)</pre> | Binary: yes, no |
| ∘ Psoriasis | Variables: eim_subcat_muco & eim_activity Derivation: 'no eim' if eim_subcat_muco≠'Psoriasis', 'Active at assessment' if eim_subcat_muco = 'Psoriasis' AND eim_activity='Active at assessment', 'Past but not active 'if eim_subcat_muco = 'Psoriasis' AND eim_activity='Past but not active' ) | Categorical: no EIM, Active at assessment, Past but not active |
| ∘ Erythema<br>nodosum | Variables: eim_subcat_muco & eim_activity Derivation: same as for Psoriasis, replacing 'Psoriasis' by 'Erythema nodosum' | |
| ∘ Pyoderma gan-<br>grenosum | Variables: eim_subcat_muco & eim_activity Derivation: same as for Psoriasis, replacing 'Psoriasis' by 'Pyoderma gangrenosum' | |
| - Aphthous stoma-<br>titis | Variables: eim_subcat_muco & eim_activity Derivation: same as for Psoriasis, replacing 'Psoriasis' by 'Aphthous stomatitis' | |
| ∘ Other | Variables: eim_subcat_muco & eim_activity Derivation: same as for Psoriasis, replacing 'Psoriasis' by ' Other' | |

|---|---|---|---|
| CTU Barra | Template: Statistical Analysis Plan (SAP) | Version: 03 | |
| CTU Bern | Code: CS_STA_TEM-11 | Valid from: 28.02.2019 | Page <b>21</b> of <b>44</b> |



| Description | Variable | Туре |
|---|---|---|
| •Musculoskeletal | eim_cat ('yes' if eim_cat='Musculoskeletal', 'no' otherwise) | |
| ∘ Inflammatory<br>arthritis | Variables: eim_subcat_muscu & eim_activity Derivation: 'no eim' if eim_subcat_muscu ≠'Inflammatory arthritis', 'Active at assessment' if eim_subcat_muscu = 'Inflammatory arthritis' AND eim_activity = 'Active at assessment', 'Past but not active ' if eim_subcat_muscu = 'Inflammatory arthritis' AND eim_activity = 'Past but not active' ) | Binary: Active at assessment, Past, but not active |
| ∘ Other | Variables: eim_subcat_muscu & eim_activity Derivation: same as for Inflammatory arthritis, replacing 'Inflammatory arthritis' by 'Other' | |
| <b>-</b> Ocular | eim_cat ('yes' if eim_cat='Ocular', 'no' otherwise) | |
| ∘ Uveitis | Variables: eim_subcat_ocular & eim_activity Derivation: 'no eim' if eim_subcat_ocular ≠ 'Uveitis', 'Active at assessment' if eim_subcat_ocular = 'Uveitis' AND eim_activity = 'Active at assessment', 'Past but not active 'if eim_subcat_ocular = 'Uveitis' AND eim_activity = 'Past but not active' ) | Binary: Active at assessment, Past, but not active |
| ∘ (Epi)scleritis | Variables: eim_subcat_ocular & eim_activity Derivation: same as for Uveitis, replacing 'Uveitis' by '(Epi)scleritis' | |
| ∘ Other | Variables: eim_subcat_ocular & eim_activity Derivation: same as for Uveitis, replacing 'Uveitis' by 'Other' | |
| •Hepatobiliary | <pre>eim_cat ('yes' if eim_cat = 'Hepatobiliary', 'no' otherwise)</pre> | |

|---|---|---|---|
| CTIL Barra | Template: Statistical Analysis Plan (SAP) | Version: 03 | |
| CTU Bern | Code: CS_STA_TEM-11 | Valid from: 28.02.2019 | Page <b>22</b> of <b>44</b> |



| Description | Variable | Туре |
|---|---|---|
| ∘ Primary<br>sclerosing<br>cholangitis | Variables: eim_subcat_hepa & eim_activity Derivation: 'no eim' if eim_subcat_hepa ≠' Primary sclerosing cholangitis', 'Active at assessment' if eim_subcat_hepa = ' Primary sclerosing cholangitis' AND eim_activity ='Active at assessment', 'Past but not active 'if eim_subcat_hepa = 'Primary sclerosing cholangiti' AND eim_activity = 'Past but not active' ) | Binary: Active at assessment, Past, but not active |
| <sup>°</sup> Cholangiocarcinoma | Variables: eim_subcat_hepa & eim_activity Derivation: same as for Primary sclerosing cholangitis, replacing 'Primary sclerosing cholangitis' by 'Cholangiocarcinoma' | |
| ∘ Primary biliary<br>cirrhosis | Variables: eim_subcat_hepa & eim_activity Derivation: same as for Primary sclerosing cholangitis, replacing 'Primary sclerosing cholangitis' by 'Primary biliary cirrhosis' | |
| - Autoimmune<br>hepatitis | Variables: eim_subcat_hepa & eim_activity Derivation: same as for Primary sclerosing cholangitis, replacing 'Primary sclerosing cholangitis' by 'Autoimmune hepatitis' | |
| ∘ Other | Variables: eim_subcat_hepa & eim_activity Derivation: same as for Primary sclerosing cholangitis, replacing 'Primary sclerosing cholangitis' by 'Other' | |
| Other UC disease ch | naracteristics | |
| Duration of disease<br>(days before base-<br>line from date of UC<br>diagnosis date | ra_uc_diag_date - ic_date | Continuous (days) |
| UC extent (location) | ra_uc_ext at baseline | Categorical: Ulcerative proctitis, Proctosig-<br>moiditis, Pancolitis, Left-sided colitis |
| CRP level | ra_crp_conc at baseline | Continuous (mg/L) |
| Full Mayo score | see data preparation 4.3 | Continuous |

|---|---|---|---|
| OTU Dama | Template: Statistical Analysis Plan (SAP) | Version: 03 | |
| CTU Bern | Code: CS_STA_TEM-11 | Valid from: 28.02.2019 | Page <b>23</b> of <b>44</b> |



| Description | Variable | Туре |
|---|---|---|
| Mayo Endoscopic subscore | ra_mayo_subscore at baseline | Categorical: Normal or inactive disease, Mild disease (erythema, decrease of vascular pattern, slight friability), Moderate disease (marked erythema, absent vascular pattern, friability, erosions), Severe disease (spontaneous bleeding, ulceration) |
| Intestinal Ultrasound at baseline | ra_ultrasound_done | Binary: Yes, No |
| fCAL at baseline | | |
| fCAL at baseline | fcal_value at baseline | Continuous |
| PRO at baseline | | |
| Stool frequency | pro_stool_freq | Categorical: Normal number of stools", 1-2 stools more than normal, 3-4 stools more than normal, 5 or more stools than normal |
| Rectal bleeding | pro_rect_bleed | Categorical: No blood seen, Blood streaks seen in stool less than half the time, Blood seen in stool most of the time, Blood alone passes |
| Urgency of defeca-<br>tion | pro_nrs_urgency | Continuous |
| Abdominal pain | pro_nrs_abd_pain | Continuous |
| Quality of sleep | pro_nrs_qual_sleep | Continuous |
| Daily fatigue | pro_nrs_fatigue | Continuous |
| Weekly fatigue | Weekly fatigue score (see data preparation 4.3) | Continuous |
| Quality of life<br>(IBDQ) | pro_ibdq_x (with x varying between 1 and 32) at baseline see data preparation 4.3 | Continuous |

# 6.5 Procedural characteristics (if applicable)

Not applicable.

### 6.6 Adherence and protocol deviations

Adherence to study protocol and to tofacitinib will not be assessed.

Main analysis will be conducted on the full analysis set (FAS). Secondary analysis will include all study participants who did not stop or interrupt the tofacitinib therapy before the week 8 visit (i.e OTAS set, see section 5.2.3).

### 6.7 Withdrawal/follow-up

Number and percentage of withdrawal and lost to follow-up will be presented in the flow chart (see section 6.3).

|---|---|---|---|
| CTO Belli | Code: CS_STA_TEM-11 | Valid from: 28.02.2019 | Page <b>24</b> of <b>44</b> |



CTU Bern

# 7. Analysis

# 7.1 Outcome definitions

Table 7-a: Derivation of study outcomes

Template: Statistical Analysis Plan (SAP)

Code: CS\_STA\_TEM-11

| Outcome | Definition | eCRF sheet | Variable | Variable<br>type | Derivation | Outcome type |
|---|---|---|---|---|---|---|
| PRIMARY OUTCOME | | | | | | - <del></del> |
| Clinical response at<br>W8 | (1) reduction in PMS from baseline of ≥2 points or (2) achieving clinical remission | PMS | PMS score (see section 4.3) pms_stool_freq pms_rect_bleed pms_glob_ass | continuous | Yes: If (PMS at W8- PMS at baseline≥2) OR PMS at W8 ≤2 AND pms_stool_freq<2 AND pms_rect_bleed<2 AND pms_glob_ass<2 at W8. | Binary:<br>Yes, no |
| SECONDARY OUTCOM | ES | I | | | | 1 |
| Clinical response at<br>W16 | (1) reduction in PMS from baseline of ≥2 points or (2) achieving clinical remission | | PMS score (see section 4.3) pms_stool_freq pms_rect_bleed pms_glob_ass | continuous | Yes: If (PMS at W16- PMS at baseline≥2) OR PMS at W16 ≤2 AND pms_stool_freq<2 AND pms_rect_bleed<2 AND pms_glob_ass<2 at W16. | Binary:<br>Yes, no |
| Clinical remission<br>W8/W16 | Clinical remission:<br>PMS of ≤ 2 with no<br>subscore >1 | | PMS score (see section 4.3) pms_stool_freq pms_rect_bleed pms_glob_ass | continuous | Yes: PMS at W8 (or 16) ≤2 AND pms_stool_freq<2<br>AND pms_rect_bleed<2 AND pms_glob_ass<2 at<br>W8 (or 16). | Binary:<br>Yes, no |
| CTU Bern SAP for: S | :<br>Study A3921395 KIC-STA | RT | Version: 1.0 | • | ] | • |

Page **25** of **44** 

Version: 03

Valid from: 28.02.2019



| Outcome | Definition | eCRF sheet | Variable | Variable type | Derivation | Outcome<br>type |
|---|---|---|---|---|---|---|
| IBDQ remission at W8/W16 | IBDQ remission: IBDQ score ≥ 170 | | IBDQ score calculated as described in section 4.3 at W8 and 16 | continuous | Yes: IBDQ at W8 (or 16) ≥170 | Binary:<br>Yes, no |
| IBDQ response at W8/W16 | IBDQ response: IBDQ score ≥16 points higher than IBDQ baseline score | | IBDQ score calculated as described in section 4.3 at baseline, W8 and 16 | continuous | Yes: IBDQ at W8 (or 16) – IBDQ at BL≥16 | Binary:<br>Yes, no |
| Biochemical remission at W8/W16 | Biochemical remission: fCAL concentration ≤250 μg/g | | fcal_value | continuous | Yes: fcal_value≤250 μg/g | Binary:<br>Yes, no |
| PROs | | | | | | |
| Stool frequency | | Stool freq, rect.<br>bleed, NRS | pro_stool_freq | Score (0-3), continuous | | Continuous |
| Rectal bleeding | | | pro_rect_bleed | Score (0-3), continuous | | Continuous |
| Urgency of defecation | | | pro_nrs_urgency | Continuous | | Continuous |
| Abdominal pain | | | pro_nrs_abd_pain | Continuous | | Continuous |
| Quality of sleep | | | pro_nrs_qual_sleep | Continuous | | Continuous |
| Daily fatigue | | | pro_nrs_fatigue | Continuous | | Continuous |
| Weekly fatigue | | FACIT-F | "pro_facit_an1", "pro_facit_an12", "pro_facit_an14"," pro_facit_an15", | Continuous | See section 4.3 | Continuous |

|---|---|---|
| | Template: Statistical Analysis Plan (SAP) | Version: 03 |
| CTU Bern | Code: CS_STA_TEM-11 | Valid from: 28 02 2019 |



| Outcome | Definition | eCRF sheet | Variable | Variable<br>type | Derivation | Outcome type |
|---|---|---|---|---|---|---|
| IBDQ<br>PMS | | PRO IBDQ<br>PMS | "pro_facit_an16", "pro_facit_an2", "pro_facit_an3", "pro_facit_an4", "pro_facit_an5", "pro_facit_an7", "pro_facit_an8", "pro_facit_hi12", "pro_facit_hi7". pro_ibdq_1 to 32 PMS score (see section 4.3) | Continuous<br>Continuous | See section 4.3 | Continuous |
| Clinical response | | fCAL | fcal_value | Continuous | | Continuous |
| EXPLORATORY OUTCO | | | | | | |
| FMS response at W8/W16. | FMS response: decrease from baseline total Mayo score of ≥3 points and ≥30%, with an accompanying decrease in the rectal bleeding subscore of ≥1 or absolute rectal bleeding subscore ≤1 | PMS & SOC<br>Assessment | ra_full_mayo (calculated as described in section 4.3) pms_rect_bleed | Continuous | | Binary:<br>Yes, no |

|----------|-----------------------------------|--------------|
|----------|-----------------------------------|--------------|

| CTIL Bown | Template: Statistical Analysis Plan (SAP) | Version: 03 | |
|---|---|---|---|
| CTU Bern | Code: CS_STA_TEM-11 | Valid from: 28.02.2019 | Page <b>27</b> of <b>44</b> |



| Outcome | Definition | eCRF sheet | Variable | Variable<br>type | Derivation | Outcome<br>type |
|---|---|---|---|---|---|---|
| remission at W8/W16 | Remission: a total Mayo score of ≤2, with no subscore >1 and a rectal bleeding subscore of 0 | PMS & SOC<br>Assessment | ra_full_mayo (cal-<br>culated as de-<br>scribed in section<br>4.3)<br>pms_stool_freq<br>pms_glob_ass | continuous | ra_full_mayo at W8/16 ≤2 AND [pms_stool_freq ≤ 1 AND pms_glob_ass ≤ 1 at W8/16 AND pms_rect_bleed at W8/16 = 0] | Binary:<br>Yes, no |
| mucosal healing at W8/W16. | Mucosal healing: a<br>Mayo endoscopic<br>subscore of ≤1 | SOC Assess-<br>ment | ra_mayo_subscore | continuous | ra_mayo_subscore at W8/16 ≤1 | Binary:<br>Yes, no |
| response according to IUS assessment at W8/W16. | According to treating physician's assessment of bowel wall thickness, normalization and extension; bowel wall vascularity, loss of stratification, loss of colonic haustration, structure formation and hyperechogenic reaction adjacent to the bowel wall. | SOC Assessment | ra_global_eval | categorical | Yes: ra_global_eval %in% c('re-sponse', 'remission') | Binary:<br>Yes, no |
| remission according to IUS assessment at W8/W16. | According to treat-<br>ing physician's as-<br>sessment of bowel<br>wall thickness, nor- | SOC Assess-<br>ment | ra_global_eval | categorical | Yes: ra_global_eval ='remission' | Binary:<br>Yes, no |

|---|---|---|
| Code: CS_STA_TEM-11 | Valid from: 28.02.2019 | Page <b>28</b> of <b>44</b> |



| Outcome | Definition | eCRF sheet | Variable | Variable<br>type | Derivation | Outcome<br>type |
|---|---|---|---|---|---|---|
| | malization and extension; bowel wall vascularity, loss of stratification, loss of colonic haustration, structure formation and hyperechogenic reaction adjacent to the bowel wall. | | | | | |
| individual improvement in EIM reported at BL at W8/W16 15 outcome/variables | EIM improvement<br>for EIM reported at<br>BL | Extra Intestinal<br>Manifestations<br>(EIM) | eim_cat eim_subcat eim_activity ('Past, but not active' vs. active at assessment) | -Categorical<br>-Categorical<br>- Binary | See section 4.3 for EIM improvement status at week_x (x can be equal to 8 or 16) Yes: EIM improvement status == Improved | Binary:<br>Yes, no |
| Categorical improvement 5 variables/outcomes | EIM improvement is reported for at least one of the subcategories of the studied category. | Extra Intestinal<br>Manifestations<br>(EIM) | eim_cat eim_activity ('Past, but not active' vs. active at assessment) | -Categorical<br>- Binary | Yes: eim_cat==the studied category AND eim_activity=='Past, but not active' | Binary:<br>Yes, no |
| Average daily dose of Tofacitinib during the trial | TORY OUTCOMES | Baseline Tofacitinib Change in Tofacitinib Exposure | | | See section 4.3 | Binary:<br><15mg<br>tofa-cit-<br>inib/day, |

|---|---|---|
| CTO Belli | Code: CS_STA_TEM-11 | Valid from: 28 02 2019 |



| ≥15 mg to- |
|--------------|
| fa- |
| citinib/day |
| Binary: ac- |
| tive UC, in- |
| active UC |
| Binary: |
| Yes, no |
| Binary: |
| Yes, no |
| , |
| Binary: |
| Yes, no |

| CTU Bern | SAP for: Study A3921395 KIC-START | 5 KIC-START Version: 1.0 |
|---|---|---|
| | 1 | |
| C TO Bern | Code: CS_STA_TEM-11 | Valid from: 28 02 2019 |



| Outcome | Definition | eCRF sheet | Variable | Variable<br>type | Derivation | Outcome type |
|---|---|---|---|---|---|---|
| Loss of colonic haustration at W8 & 16 | | SOC Assess-<br>ment, Intestinal<br>Ultrasound | ra_loss_col_haus | | | Binary:<br>Yes, no |
| Structure formation at W8 & 16 | | SOC Assess-<br>ment, Intestinal<br>Ultrasound | ra_struct_form | | | Binary:<br>Yes, no |
| Hyperechogenic reaction adjacent to the bowel wall | | SOC Assess-<br>ment, Intestinal<br>Ultrasound | ra_hyper_react | | | Binary:<br>Yes, no |
| Occurrence of new EIM at W8/W16 15 outcome/variables | Occurrence of<br>EIM not reported<br>at BL | Extra Intestinal<br>Manifestations<br>(EIM) | eim_cat eim_subcat eim_activity ('Past, but not active' vs. active at assessment) | -Categorical<br>-Categorical<br>- Binary | See section 4.3 for EIM improvement status at week_x (x can be equal to 8 or 16) Yes: EIM improvement status == New occurrence | Binary:<br>Yes, no |
| Number of EIMs at<br>W8 and 16 | | Extra Intestinal<br>Manifestations<br>(EIM) | | | See section 4.3 | Continuous |
| Number of comorbidities at W8 and 16 | | Extra Intestinal<br>Manifestations<br>(EIM) | | | See section 4.3 | Continuous |
| PMS stool frequency subscore | | PMS | | | See section 4.3 | Continuous |
| PMS rectal bleeding subscore | | PMS | | | See section 4.3 | Continuous |

|---|---|---|---|
| OTU B | Template: Statistical Analysis Plan (SAP) | Version: 03 | |
| CTU Bern | Code: CS_STA_TEM-11 | Valid from: 28.02.2019 | Page <b>31</b> of <b>44</b> |



| Outcome | Definition | eCRF sheet | Variable | Variable<br>type | Derivation | Outcome<br>type |
|---|---|---|---|---|---|---|
| PMS physician's global assessment subscore | | PMS | | | See section 4.3 | Continuous |

|---|---|---|---|
| OTU D | Template: Statistical Analysis Plan (SAP) | Version: 03 | |
| CTU Bern | Code: CS_STA_TEM-11 | Valid from: 28.02.2019 | Page <b>32</b> of <b>44</b> |



Table 7-b: EIM categories and subcategories

| Variable | Category | Subcategory |
|---|---|---|
| Hepatobiliary; Primary sclerosing cholangitis | Hepatobiliary | Primary sclerosing cholangitis |
| Hepatobiliary; Cholangiocarcinoma | | Cholangiocarcinoma |
| Hepatobiliary; Primary biliary cirrhosis | | Primary biliary cirrhosis |
| Hepatobiliary; Autoimmune hepatitis | | Autoimmune hepatitis |
| Hepatobiliary; Other | | Other |
| Ocular; Uveitis | Ocular | Uveitis |
| Ocular; (Epi)scleritis | | (Epi)scleritis |
| Ocular; Other | | Other |
| Musculoskeletal; Inflammatory arthritis | Musculoskeletal | Inflammatory arthritis |
| Musculoskeletal; Other | | Other |
| Mucocutaneous; Psoriasis | Mucocutaneous | Psoriasis |
| Mucocutaneous; Erythema nodosum | | Erythema nodosum |
| Mucocutaneous; Pyoderma gangrenosum | | Pyoderma gangrenosum |
| Mucocutaneous; Aphthous stomatitis | | Aphthous stomatitis |
| Other; Other | Other | Other |

|---|---|---|---|
| OTU Dama | Template: Statistical Analysis Plan (SAP) | Version: 03 | |
| CTU Bern | Code: CS STA TEM-11 | Valid from: 28.02.2019 | Page <b>33</b> of <b>44</b> |



### 7.2 Analysis methods

#### 7.2.1 Primary analysis

In the primary analysis, all patients will be analyzed using the FAS set.

Proportions of patients achieving clinical, IBDQ and biochemical response and remission at W8 and W16 will be calculated and reported with the associated 95% Wilson confidence interval.

The course of continuous secondary outcomes (PMS, IBDQ score, PROs and fCAL) and of the exploratory additional PMS subscore outcomes over time will be depicted by box plots showing medians, quartiles, and outlying values. For these outcomes and for Medians and associated quartiles at baseline, W8, and W16 will be reported in a table.

For these outcomes, the change from baseline will be calculated at each time point as the observed value minus the value measured at baseline. The course of change over time, will be depicted by box plots showing medians, quartiles, and outlying values. Medians and associated quartiles at W8 and W16 will be reported in a table.

The course of fCAL over time will be shown separately for patients with and without clinical response as well as for patients with and without remission at W8 and W16. Medians and associated quartiles at W8 and W16 will be reported in a table.

Correlation between PRO outcomes and PMS, PMS subscores, IBDQ score and fCAL concentrations will be assessed at BL, W8 and W16 by the Spearman correlation coefficient. For each time point the correlation coefficient will be presented in a table.

Average daily dose of Tofacitinib during the trial, active UC and others additional outcomes assessed via ultrasound, number of comorbidities and EIM number, improvement, and new occurrence will be described at W8 and 16 in descriptive tables. Categorical variables will be summarized as number and proportion, continuous variables as median with quartiles range or mean with standard deviation, as appropriate.

#### 7.2.2 Secondary analyses

If more than 2 patients are excluded from the on-tofacitinib analysis set (OTAS), all analysis described in the primary analysis section above will be conducted on the OTAS population.

#### 7.2.3 Sensitivity analyses

Code: CS STA TEM-11

Not applicable.

|-----------|-------------------------------------------|--------------|
| CTII Bern | Template: Statistical Analysis Plan (SAP) | Version: 03 |

Valid from: 28.02.2019




UNIVERSITÄT

Faculty of Medicine
CTU Bern

### 7.2.4 Subgroup analyses

Not applicable.

#### 7.2.5 Additional analyses

Not applicable.

#### 7.3 Interim analyses

Not applicable.

### 7.4 Missing data

Missing data will be ignored.

Rules for calculations of the different scores in the presence of missing information are detailed in the above sections.

# 7.5 Safety evaluation

Safety data are collected for the purpose of meeting routine pharmacovigilance reporting requirements. Safety data will not be analyzed, but number and frequency of (S)AEs will be reported, including tabulations by severity, number of withdrawals or does reductions due to AE, and by system organ class (SOC).

#### 7.6 Subproject (if applicable)

Not applicable.

#### 7.7 Statistical software

All the analysis will be done using R (version 3.6.0 or higher) [16].

### 7.8 Quality control

A second statistician will reproduce the primary analysis based on the exported data. If results deviate, the reason for the difference will be determined and a consensus must be reached.

# 8. Presentation of the results - Tables, Listings and Figures

# 8.1 Figures

#### 8.1.1 Flow chart

See section 6.3.

|---|---|---|---|
| CTU Barra | Template: Statistical Analysis Plan (SAP) | Version: 03 | |
| CTU Bern | Code: CS STA TEM-11 | Valid from: 28.02.2019 | Page <b>35</b> of <b>44</b> |




CTU Bern

8.1.2 Course of the PMS, PROs and fCAL concentration.

Figure (10 subplots): Boxplot showing the course of the PMS, PROs (each component separately) and fCAL concentration.

Figure (4 subplots): Boxplot (or line plot) showing the course of fCAL for patients with (subplot A) and without (subplot B) clinical response as well as for patients with (subplot C) and without (subplot D) remission at week 8 and 16.

#### 8.2 Tables

# 8.2.1 Study participants

Baseline characteristics presented in the baseline table of this document (see section 6.4) will be presented in different tables presenting the:

table a. Key baseline characteristics including:

- Patient demographics,
- o Concomitant medication at baseline,
- o UC medication,
- Main UC disease characteristics.
- UC treatment history excluding prior exposure to oral & topical aminosalicylates, locally acting & systemic cortico-steroids (e.g. budesonide, prednisone), Thiopurines (e.g. AZA, 6-MP), Other immunosuppressants (e.g. cyclosporine, tacrolimus), TNF inhibitors (TNFi),
- fCAL at baseline,
- o PRO at baseline,

Code: CS STA TEM-11

o Co-morbidities

table b. EIMs table c. SOC IUS

CTU Bern

In each of these tables, categorical variables will be summarized as number and proportion, continuous variables as median with quartiles range or mean with standard deviation, as appropriate.

Prior exposure to oral & topical aminosalicylates, Locally acting & systemic corticosteroids (e.g. budesonide, prednisone), Thiopurines (e.g. AZA, 6-MP), Other immunosuppressants (e.g. cyclosporine, tacrolimus), TNF inhibitors (TNFi) will be presented as number and percentage in a separate table as below.

Table c: UC treatment history: Summary of primary reason for discontinuation of prior UC therapies by treatment group

| Prior UC therapy, n (%) | ' ' | Intolerance/side<br>effects | Unknown |
|---|---|---|---|
| Oral & topical aminosalicylates | | | |

|---|---|
| Template: Statistical Analysis Plan (SAP) | Version: 03 |

Valid from: 28.02.2019



Faculty of Medicine
CTU Bern

| Prior UC therapy, n (%) | • | Lack of/ insufficient response | Intolerance/side<br>effects | Unknown |
|---|---|---|---|---|
| Localized/Topical corticosteroids (e.g. budesonide) | | | | |
| Systemic corticosteroids (e.g. prednisone) | | | | |
| Thiopurines (e.g. AZA, 6-MP) | | | | |
| Other immunosuppressants (e.g. cyclosporine, tacrolimus) | | | | |
| TNF inhibitors (TNFi) | | | | |
| Vedolizumab | | | | |
| Ustekinumab | | | | |

# 8.2.2 Efficacy Outcomes at W8 and W16

Legend:

| Primary outcome |
|----------------------|
| Secondary outcomes |
| Exploratory outcomes |

### a. Main outcomes

| Outcome | Proportion (%) of outcomes (n/N) [95% CI] * | |
|---|---|---|
| | W8 | W16 |
| Clinical response | % (n/N) [CI] | % (n/N) [CI] |
| Clinical remission | % (n/N) [CI] | % (n/N) [CI] |
| IBDQ response | % (n/N) [CI] | % (n/N) [CI] |
| IBDQ remission | % (n/N) [CI] | % (n/N) [CI] |
| Biochemical remission | % (n/N) [CI] | % (n/N) [CI] |
| FMS response | % (n/N) [CI] | % (n/N) [CI] |
| Remission | % (n/N) [CI] | % (n/N) [CI] |
| Mucosal healing | % (n/N) [CI] | % (n/N) [CI] |
| Response according to IUS assessment | % (n/N) [CI] | % (n/N) [CI] |
| Remission according to IUS assessment | % (n/N) [CI] | % (n/N) [CI] |
| Individual improvement in EIM | % (n/N) [CI] | % (n/N) [CI] |
| Categorical improvement in EIM | % (n/N) [CI] | % (n/N) [CI] |

# Footnotes:

|----------|-----------------------------------|--------------|

|---|---|---|---|
| CTO Bern | Code: CS_STA_TEM-11 | Valid from: 28.02.2019 | Page <b>37</b> of <b>44</b> |



UNIVERSITÄT

Faculty of Medicine
CTU Bern

\* 95% Wilson confidence interval

Definitions for clinical response, clinical remission, IBDQ response, IBDQ remission, Biochemical remission, FMS response, remission, mucosal healing, response according to IUS assessment, remission according to IUS assessment, improvement in EIM.

- \*\*Results presented for each EIM and EIM category
- \*\*\* Result presented for ascending colon, transverse colon, descending colon and sigmoid colon.

#### 8.2.3 Temporal variation of PMS, PROs and fCAL concentration

Value and change from baseline at baseline, W8 and W16 of PMS, PROs (each component separately) and fCAL concentration (values presented as median and quartiles).

| | Outcome | | Value at | | | ge from<br>line at |
|---|---|---|---|---|---|---|
| Category | Name | Baseline | W8 | W16 | W8 | W16 |
| | | Median | Median | Median | Median | Median |
| PRO | Stool frequency | [Q1;Q3] | [Q1;Q3] | [Q1;Q3] | [Q1;Q3] | [Q1;Q3] |
| PRO | Rectal bleeding | | | | | |
| PRO | Urgency of defecation | | | | | |
| PRO | Abdominal pain | | | | | |
| PRO | Quality of sleep | | | | | |
| PRO | Daily fatigue | | | | | |
| PRO | Weekly fatigue | | | | | |
| PRO | Quality of life (IBDQ) | | | | | |
| PMS | PMS | | | | | |
| fCAL | fCAL concentration | | | | | |

# 8.2.3.1 Temporal variation of the fcal concentration in patients with and without clinical response and remission

Value and change from baseline at baseline, W8 and W16 of fCAL concentration stratified by clinical outcomes at W8 and W16. (Values presented as median and quartiles)

| Outcome | Value at | | | Change from<br>baseline at | |
|---------|----------|----|-----|----------------------------|-----|
| | Baseline | W8 | W16 | W8 | W16 |

fCAL all patients

fCAL for patients with clinical response at W8

fCAL for patients without clinical response W8

fCAL for patients with clinical response at W16

|---|---|---|
| CTIL Dawn | Template: Statistical Analysis Plan (SAP) | Version: 03 |
| CTU Bern | Code: CS_STA_TEM_11 | Valid from: 28 02 2019 |



UNIVERSITÄT

Faculty of Medicine
CTU Bern

fCAL for patients without clinical response W16

fCAL for patients with clinical remission at W8

fCAL for patients without clinical remission W8

fCAL for patients with clinical remission at W16

fCAL for patients without clinical remission W16

Footnote: Definitions for clinical response and clinical remission according to IUS assessment.

|---|---|---|
| | Tarrallatas Chatistical Amalusia Plan (CAP) | V |
| O I O DCIII | Code: CS_STA_TEM-11 | Valid from: 28 02 2010 |



# 8.3 Correlation between PRO and PMS, IBDQ score and fCAL concentrations outcomes.

Correlations measures (Spearman correlation coefficients) will be assessed at BL (Table a), W8 (Table b) and W16 (Table c). Results will be presented in similar but separated tables.

| | Stool<br>frequ<br>ency | Rect<br>al<br>blee<br>ding | Urge<br>ncy<br>of<br>defec<br>ation | Abdo<br>minal<br>pain | Qu<br>alit<br>y of<br>sle<br>ep | Dai<br>ly<br>fati<br>gu<br>e | We<br>ekly<br>fati<br>gue | Qu<br>alit<br>y of<br>life<br>(IB<br>DQ | P<br>M<br>S | PM<br>S<br>sub<br>-<br>sco<br>re1 | PM<br>S<br>sub<br>-<br>sco<br>re2 | PM<br>S<br>sub<br>-<br>sco<br>re3 | fC<br>A<br>L |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Stool | | | | | | | | | | | | | |
| frequency | | | | | | | | | | | | | |
| Rectal bleeding | | | | | | | | | | | | | |
| Urgency of defecation | | | | | | | | | | | | | |
| Abdominal pain | | | | | | | | | | | | | |
| Quality of sleep | | | | | | | | | | | | | |
| Daily fatigue | | | | | | | | | | | | | |
| Weekly | | | | | | | | | | | | | |
| fatigue | | | | | | | | | | | | | |
| Quality of life<br>(IBDQ) | | | | | | | | | | | | | |
| PMS | | | | | | | | | | | | | |
| Stool fre-<br>quency<br>subscore<br>of PMS | | | | | | | | | | | | | |
| Rectal<br>bleeding<br>subscore<br>of PMS | | | | | | | | | | | | | |
| PGA sub-<br>score of<br>PMS | | | | | | | | | | | | | |
| fCAL | | | • | | | | | | | | | | |

|---|---|
| Templete: Statistical Applyais Plan (SAD) | Version: 03 |



# 8.4 Additional exploratory outcomes

Additional exploratory outcomes listed in section 7.1 will be presented at W8 and 16 in separate descriptive tables. In each of these tables, categorical variables will be summarized as number and proportion, continuous variables as median with quartiles range or mean with standard deviation, as appropriate.

| | W8 | W16 |
|---|---|---|
| Average daily dose of Tofacitinib during the trial | median [Q1, Q3], or mean (sd) | median [Q1, Q3], or mean (sd) |
| Active UC at W8 and 16 based on IUS assessments | % (n/N) [CI] | % (n/N) [CI] |
| Extension of wall-thickening* | % (n/N) [CI] | % (n/N) [CI] |
| Normalization of wall-thickening* | % (n/N) [CI] | % (n/N) [CI] |
| Loss of stratification | % (n/N) [CI] | % (n/N) [CI] |
| Loss of colonic haustration | % (n/N) [CI] | % (n/N) [CI] |
| Structure formation | % (n/N) [CI] | % (n/N) [CI] |
| Hyperechogenic reaction adjacent to the bowel wall | % (n/N) [CI] | % (n/N) [CI] |
| Occurrence of new EIM | % (n/N) [CI] | % (n/N) [CI] |
| Number of EIMs | median [Q1, Q3], or mean (sd) | median [Q1, Q3], or mean (sd) |
| Number of comorbidities | median [Q1, Q3], or mean (sd) | median [Q1, Q3], or mean (sd) |
| PMS stool frequency subscore | median [Q1, Q3], or mean (sd) | median [Q1, Q3], or mean (sd) |
| PMS rectal bleeding subscore | median [Q1, Q3], or mean (sd) | median [Q1, Q3], or mean (sd) |
| PMS physician's global assess-<br>ment subscore | median [Q1, Q3], or mean (sd) | median [Q1, Q3], or mean (sd) |

<sup>\*</sup> For Ascending, descending, Sigmoid and transverse colon

|---|---|---|---|
| | T | N | |
| C 10 Delli | Code: CS_STA_TEM-11 | Valid from: 28 02 2019 | Page <b>41</b> of <b>4</b> 4 |



UNIVERSITÄT

Faculty of Medicine
CTU Bern

# 8.5 Safety Data

# 8.5.1 Summary of AEs

| | All Causalities | Treatment Related |
|---|---|---|
| Number of AEs | | |
| Subjects with AEs [n (%)] | | |
| Subjects with SAEs <sup>a</sup> [n (%)] | | |
| Subjects with severe AEsb [n (%)] | | |
| Subjects permanently with-<br>drawn from tofocitinib due to<br>AEsc [n (%)] | | |
| Subjects with tofacitinib dose reduced or temporary discontinuation tofacitinib due to AEs [n (%)] | | |

#### Footnotes:

Included events from study database, even those that occurred after discontinuation of drug under study. Except for the number of AEs, subjects were counted only once per treatment in each row.

- <sup>a</sup> SAEs were determined according to the investigator's assessment.
- b. Severity counts were based on the maximum severity or grade of events.
- <sup>c.</sup> Discontinuation of tofacitinib due to AE based on the AE CRF is summarized, and numbers shown include subjects withdrawn for an AE of UC.

# 8.5.2 Severity of AEs, by system organ class and preferred term

| System organ | n (%) | Mild | Moderate | Severe |
|--------------|-------|------|----------|--------|
| class | | | | |
| Preferred | | | | |
| Term | | | | |
| SOC 1 | | | | |
| PTi | | | | |
| SOC 2 | | | | |
| PTi | | | | |
| PTi+1 | | | | |

|---|--------------|
| T | \/i00 |

| CTU Davis | Template: Statistical Analysis Plan (SAP) | Version: 03 | |
|---|---|---|---|
| CTU Bern | Code: CS_STA_TEM-11 | Valid from: 28.02.2019 | Page <b>42</b> of <b>44</b> |



Faculty of Medicine

CTU Bern

# 9. Changes from the protocol

Table x: Changes from protocol

| Header | Change | Reason |
|---|---|---|
| N patients | Sample size | Following Pfizer internal decision, recruitment was prematurely stopped after the enrollment of 18 patients. |
| Addition of new exploratory outcomes | <ul> <li>Average daily dose of Tofacitinib during the trial</li> <li>Active UC at W8 and W16</li> <li>Normalization of wall-thickening,</li> <li>Loss of stratification at W8 &amp; W16,</li> <li>Loss of colonic haustration at W8 &amp; W16,</li> <li>Structure formation at W8 &amp; W16,</li> <li>Hyperechogenic reaction adjacent to the bowel wall,</li> <li>Occurrence of new EIM at W8/W16,</li> <li>Number of EIMs at W8 and W16,</li> <li>Number of comorbidities at W8 and W16,</li> <li>PMS stool frequency subscore,</li> <li>PMS rectal bleeding subscore,</li> <li>PMS physician's global assessment subscore</li> </ul> | Sponsor decision |
| PPset | No analysis will be conducted on the PPset | Only 18 patients were recruited |
| Secondary analysis | - The effect of participants' baseline characteristics on change in PMS, PROs and fCAL values will not be assessed - subgroup analysis will not be conducted | Only 18 patients were recruited |

|---|---|---|
| Code: CS_STA_TEM-11 | Valid from: 28.02.2019 | Page <b>43</b> of <b>44</b> |



#### 10. References

- 1. Lair-Mehiri, L., et al., Real-world evidence of tofacitinib effectiveness and safety in patients with refractory ulcerative colitis. Dig Liver Dis, 2020. **52**(3): p. 268-273.
- 2. Biemans, V.B.C., et al., *Tofacitinib for ulcerative colitis: results of the prospective Dutch Initiative on Crohn and Colitis (ICC) registry.* Aliment Pharmacol Ther, 2020. **51**(9): p. 880-888.
- 3. Hoffmann, P., et al., *Tofacitinib in Treatment-Refractory Moderate to Severe Ulcerative Colitis:* Real-World Experience from a Retrospective Multicenter Observational Study. J Clin Med, 2020. **9**(7).
- 4. Honap, S., et al., Real-world Effectiveness of Tofacitinib for Moderate to Severe Ulcerative Colitis: A Multicentre UK Experience. J Crohns Colitis, 2020. **14**(10): p. 1385-1393.
- 5. Shimizu, H., et al., Rapid prediction of 1-year efficacy of tofacitinib for treating refractory ulcerative colitis. Intest Res, 2021. **19**(1): p. 115-118.
- 6. Weisshof, R., et al., Real-World Experience with Tofacitinib in IBD at a Tertiary Center. Dig Dis Sci, 2019. **64**(7): p. 1945-1951.
- 7. Chaparro, M., et al., *Tofacitinib in Ulcerative Colitis: Real-world Evidence From the ENEIDA Registry*. J Crohns Colitis, 2021. **15**(1): p. 35-42.
- 8. Deepak, P., et al., Safety of Tofacitinib in a Real-World Cohort of Patients With Ulcerative Colitis. Clin Gastroenterol Hepatol, 2020.
- 9. Opheim, R., et al., Fatigue interference with daily living among patients with inflammatory bowel disease. Qual Life Res, 2014. **23**(2): p. 707-17.
- 10. Farrell, D., G. McCarthy, and E. Savage, *Self-reported Symptom Burden in Individuals with Inflammatory Bowel Disease.* J Crohns Colitis, 2016. **10**(3): p. 315-22.
- 11. Sandborn, W.J., et al., Correlation Between Concentrations of Fecal Calprotectin and Outcomes of Patients With Ulcerative Colitis in a Phase 2 Trial. Gastroenterology, 2016. **150**(1): p. 96-102.
- 12. Kieser, M., *Methods and Applications of Sample Size Calculation and Recalculation in Clinical Trials*. 2020: Springer International Publishing.
- 13. SOP Statistical data validation, CS\_STA\_SOP\_02, version 03, 11.09.2018.
- 14. SwissMedic. Xeljanz®: Information for Healthcare Professionals. [cited 2018 April 30]; Prod. Inf.]. Available from: <a href="https://www.swissmedicinfo.ch">www.swissmedicinfo.ch</a>.
- 15. http://www.consort-statement.org/consort-2010.
- 16. R Core Team, R: A Language and Environment for Statistical Computing. 2019.

|---|---|---|
| Code: CS_STA_TEM-11 | Valid from: 28.02.2019 | Page <b>44</b> of <b>44</b> |